CLINICAL TRIAL: NCT04931615
Title: The Influence of ARTISS on Post-operative Abdominal Drainage and Seroma Formation in DIEP/MS-TRAM Free Flap Breast Reconstruction Patients
Brief Title: ARTISS a Single-centre Randomised Control Study
Acronym: ARTISS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mid and South Essex NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 287482; 2021-002624-20 (EudraCT Number)
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2023-10

CONDITIONS: Breast Neoplasms; Mammaplasty
Keywords: muscle-sparing transverse rectus abdominis myocutaneous flap; Deep Inferior Epigastric Artery Perforator
MeSH Terms: conditions — Breast Neoplasms | interventions — Freezing

STUDY DESIGN:
Intervention Model Description: Randomised controlled trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Blinded patient and blinded assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- without ARTISS (Placebo Comparator): Surgery performed without active comparative
  Interventions: Other: no ARTISS
- with ARTISS (Active Comparator): Surgery performed with active comparative
  Interventions: Drug: ARTISS 4mL Fibrin Sealant Topical Solution (Frozen)

INTERVENTIONS:
Drug: ARTISS 4mL Fibrin Sealant Topical Solution (Frozen) — Wound sealant
  Arms: with ARTISS
Other: no ARTISS — Wound closed without sealant
  Arms: without ARTISS

SUMMARY:
The Influence of ARTISS on post-operative abdominal drainage and seroma formation in DIEP/MS-TRAM free flap breast reconstruction patients.

DETAILED DESCRIPTION:
The principle aim of the study is to investigate the effect of ARTISS on abdominal wound drainage whether this could result in earlier drain removal and earlier patient discharge from hospital. The primary outcome investigated will be post- operative abdominal drainage duration in days which is vital information during this Covid pandemic to reduce hospital stay (and therefore possible Covid exposure) which could result in earlier discharge from hospital, as well as significantly reducing cost of the procedure to the NHS and frees in-patient beds for more efficient use of resources.

ELIGIBILITY:
Inclusion Criteria:

* Female adult (age 18-80)
* Patients planned for immediate or delayed DIEP/MS-TRAM breast reconstruction

Exclusion Criteria:

* Patients who are unable to consent or do not consent
* Clotting disorder
* Pregnancy
* Individuals whose immune system is depressed or who have some types of anaemia (e.g. sickle cell disease or haemolytic anaemia).
* COVID positive
* Known previous allergic reactions to ARTISS

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
post-operative abdominal mean drainage duration | 42 days
  post-operative abdominal mean drainage duration

CONTACTS AND LOCATIONS:
Overall Officials: Mary Morgan, MD, Study Chair — Mid and South Essex NHS Foundation Trust
Locations (1):
- Mid and South Essex NHS Foundation Trust, Broomfield, Essex, United Kingdom